CLINICAL TRIAL: NCT00376571
Title: Nordic Bifurcation Study. How to Use Drug Eluting Stents (DES) in Bifurcation Lesions? A Strategy of Routine Stenting Both Main Vessel and Side Branch Versus a Strategy of Routine Main Vessel Stenting and Optional Treatment of Side Branch
Brief Title: Nordic Bifurcation Study. How to Use Drug Eluting Stents (DES) in Bifurcation Lesions?
Acronym: BIFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040136
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: PCI; Bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stenting of main vessel and side branch (Experimental): Percutaneous coronary intervention
  Interventions: Procedure: Percutaneous coronary intervention
- No side branch treatment (Experimental): Percutaneous coronary intervention
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Comparing treatment of either "no side branch treatment" versus "stenting of main vessel and side branch treatment"
  Other Names: PCI; PTCA

SUMMARY:
How to use drug eluting stents (DES) in bifurcation lesions. A strategy of routine stenting of both main vessel and side branch versus a strategy of routine main vessel stenting and optional treatment of side branch. A randomized Nordic multicenter study including 400 patients with angina pectoris with clinical angiographic follow-up.

DETAILED DESCRIPTION:
Design:

* Randomized open multicentre trial.

Patients:

* Number 400.

Inclusion criteria:

* Stable or unstable AP.
* Bifurcation lesion of "LAD/diagonal", "Cx/obtuse marginal", "RCA-PDA/posterolateral branch or LM/Cx/LAD in a right dominant system.
* Diameter of main vessel by visual estimate > 2.5 mm.
* Diameter of side branch by visual estimate > 2.0 mm.
* Signed informed consent.

Exclusion criteria:

* ST-elevation Acute Myocardial infarction (AMI) within 24 hours.
* Expected survival > 1 year.
* S-creatinine > 200 Umol/l.
* Allergy to Aspirin, Clopidogrel or Ticlopidine.
* Allergy to sirolimus/paclitaxel.
* Left main bifurcation in a non-right dominant system.

Randomization:

* Treatment strategy routine stenting of both main vessel and side branch versus routine main vessel stenting and optional treatment of side branch.

Primary end-point:

* Combined end-point of cardiac death, myocardial infarction, stent thrombosis or TVR after 6 months.

Secondary end-point:

* Clinical

  1 MACE (cardiac death, myocardial infarction, stent thrombosis or TVR) during hospital period, after 1 and 8 months.

  2 Cardiac death during hospital period, after 1, 6 and 8 months. 3 Myocardial infarction during hospital period, after 1, 6 and 8 months. 4 Stent thrombosis during hospital period, after 1, 6 and 8 months. 5 TVR during hospital period, after 1, 6 and 8 months. 6 Total death during hospital period, after 1, 6 and 8 months. 7 TLR during hospital period, after 1, 6 and 8 months. 8 Myocardial infarction related to index procedure. 9 CCS angina score after 6 and 8 months.
* Angiographic

  1. Angiographic restenosis (>50% diameter stenosis)of main vessel and occlusion of side branch
  2. Late loss of main vessel and side branch after 8 months.
  3. Percentual diameter stenosis of main vessel and side branch after 8 months.
  4. Angiographic restenosis (>50% diameter stenosis) rate of main vessel and side branch after 8 months.

End-point evaluation:

Primary and secondary end-points will be assessed by an independent end-point committee. The end-point committee will consist of experienced interventional cardiologists. Detailed end-point definitions:

* Q-wave myocardial infarction: Appearance of a new Q-wave in two or more contiguous leads on ECG.
* Non-Q-wave myocardial infarction: Infarction, which is considered present in a patient having clinical, angiographic, electrocardiographic and/or laboratory evidence of myocardial necrosis with an ECG showing no new Q-waves.
* Procedure related myocardial infarction: A threefold increase or CK-MB or Troponin-T/I.
* Target lesion revascularization: Coronary bypass operation with grafting or PCI of index lesion.
* Target vessel revascularization: Coronary bypass operation with grafting or PCI of index vessel.
* Stent thrombosis: Thrombotic occlusion of index stent/stents.
* Vessel measurement:

  1 Proximal reference diameter: Vessel diameter proximal to lesion. 2 Distal reference diameter: Vessel diameter distal to lesion. 3 Reference diameter: Mean of proximal and distal vessel diameter. 4 Percentual diameter stenosis: (Reference diameter - minimal luminal diameter)/reference diameter in percent.
* Angiographic restenosis: > 50% diameter stenosis.

Angiographic core lab:

The index and the follow-up angiograms will be assessed blindly at the QCA core lab. at Department of Cardiology, Skejby Hospital, DK-8200 Aarhus N, Denmark.

* Definition of index angiography: The angiography obtained during the PCI procedure will be used as index angiography.

* Definition of follow-up angiography: After 8 months a conventional diagnostic angiography will be performed and the projections used at the index angiography will be repeated.

Steering committee:

The steering committee will consist of one or two investigators from each center. All steering committee members will have full access to the database and will participate in the interpretation of data.

Progress of the study:

The progress of the study will be checked on a weekly basis by the steering committee. They will receive and evaluate data on inclusion rate and the primary end-point event rate. Further, the steering committee will receive and evaluate the weekly safety data on the rate of stent thrombosis in the two groups.

Statistics and data management:

* The statistical analyses will be performed by UNI-C, University of Aarhus.
* Primary end-point: The composite of the primary end-point at 6 months follow-up will be analyzed by the Kaplan-Meier method. Differences between the event-free survival curves will be compared with the use of the Wilcoxon and log-rank tests. Two-sided test is used and the p-value considered to indicate significance will be 0.05.
* Secondary end-points and other parameters: For continuous variables, differences between the treatment groups will be evaluated by analysis of variance or Wilcoxon's rank-sum test. For discrete variables, differences will be expressed as counts and percentages will be analyzed with Fisher's exact test. Secondary end-points will be assessed after 8 months. Two-sided test is used and the p-value considered to indicate significance will be 0.05.

Safety:

* For safety reasons, stent thrombosis after one month will be monitored continuously. A stent thrombosis rate of >5% in any of the treatment groups will necessitate premature termination of the trial.

Analysis population:

* Results are analyzed according to the intention-to-treat principle, i.e. patients randomized to a certain group will be followed and assessed irrespectively of the actual treatment. Protocol violations will be noted and the responsible centers notified.

Sample size calculation:

* With an expected primary end-point event rate of 30% in the "stenting main vessel and side branch group", an alpha of 5% and a power of 80%, a reduction of primary end-point event rate to 15% in the "optional side branch treatment group" can be detected with 200 patients in each group.

Randomization procedure:

* The patient will be randomized at the beginning of the PCI procedure and before any insertion of wire or balloons.
* There will be a block randomization according to centre and a stratification according to sex, age>70 years, diabetes, use of GPIIb/IIIa blocker and +/- angiographic follow-up.
* The patients will be computer randomized by a 24 hour telephone service. The PARAVOX system will be used.

Monitoring of the study:

Data will be monitored according to the GCP rules by independent professionals. During the trial, the monitor will have regular contacts with the trial site(s), including visits to ensure that the trial is conducted and documented properly in compliance with the protocol, GCP and applicable regulatory requirements.

Publication:

* Results will be published in an international cardiovascular journal. Publication and author issues will be decided by the steering committee on basis of general involvement in the study (core lab. function, end-point committee membership ect.) and of number of included patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable AP.
* Bifurcation lesion of "LAD/diagonal", "Cx/obtuse marginal", "RCA-PDA/posterolateral branch or LM/Cx/LAD in a right dominant system.
* Diameter of main vessel by visual estimate > 2.5 mm.
* Diameter of side branch by visual estimate > 2.0 mm.
* Signed informed consent.

Exclusion Criteria:

* ST-elevation AMI within 24 hours.
* Expected survival < 1 year.
* S-creatinine > 200 Umol/l.
* Allergy to Aspirin, Clopidogrel or Ticlopidine.
* Allergy to sirolimus/paclitaxel.
* Left main bifurcation in a non-right dominant system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Combined end-point of cardiac death, MI, stent thrombosis or TVR. | After 6 months

SECONDARY OUTCOMES:
Clinical: MACE (cardiac death, MI, stent thrombosis or TVR) during hospital period, after 1 and 8 months. Cardiac death, myocardial infarction, stent thrombosis, TVR, total death, TLR during hospital period, after 1, 6 and 8 months. Myocardial infarction | During hospital period, after 1, 6 and months.
Angiographic: Restenosis of the main vessel and/or occlusion of the side branch. Late loss of main vessel and side branch after 8 months. Angiographic restenosis (>50% diameter stenosis) rate of main vessel and side branch after 8 months. | After 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Leif Thuesen, MD, Study Director — Director, Cardiac Cath. Lab., Skejby Hospital, University of Aarhus
Locations (1):
- Skejby Hospital, University of Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Behan MW, Holm NR, de Belder AJ, Cockburn J, Erglis A, Curzen NP, Niemela M, Oldroyd KG, Kervinen K, Kumsars I, Gunnes P, Stables RH, Maeng M, Ravkilde J, Jensen JS, Christiansen EH, Cooter N, Steigen TK, Vikman S, Thuesen L, Lassen JF, Hildick-Smith D. Coronary bifurcation lesions treated with simple or complex stenting: 5-year survival from patient-level pooled analysis of the Nordic Bifurcation Study and the British Bifurcation Coronary Study. Eur Heart J. 2016 Jun 21;37(24):1923-8. doi: 10.1093/eurheartj/ehw170. Epub 2016 May 8. PMID 27161619
- [Derived] Kervinen K, Niemela M, Romppanen H, Erglis A, Kumsars I, Maeng M, Holm NR, Lassen JF, Gunnes P, Stavnes S, Jensen JS, Galloe A, Narbute I, Sondore D, Christiansen EH, Ravkilde J, Steigen TK, Mannsverk J, Thayssen P, Hansen KN, Helqvist S, Vikman S, Wiseth R, Aaroe J, Jokelainen J, Thuesen L; Nordic PCI Study Group. Clinical outcome after crush versus culotte stenting of coronary artery bifurcation lesions: the Nordic Stent Technique Study 36-month follow-up results. JACC Cardiovasc Interv. 2013 Nov;6(11):1160-5. doi: 10.1016/j.jcin.2013.06.009. PMID 24262616
- [Derived] Behan MW, Holm NR, Curzen NP, Erglis A, Stables RH, de Belder AJ, Niemela M, Cooter N, Chew DP, Steigen TK, Oldroyd KG, Jensen JS, Lassen JF, Thuesen L, Hildick-Smith D. Simple or complex stenting for bifurcation coronary lesions: a patient-level pooled-analysis of the Nordic Bifurcation Study and the British Bifurcation Coronary Study. Circ Cardiovasc Interv. 2011 Feb 1;4(1):57-64. doi: 10.1161/CIRCINTERVENTIONS.110.958512. Epub 2011 Jan 4. PMID 21205942